CLINICAL TRIAL: NCT06506578
Title: Characterization of Nausea Induced by Radiation of the Dorsal Vagal Complex in the Context of Benign Brain Tumors (NausiCAA)
Brief Title: Nausea Induced by Radiation of the Dorsal Vagal Complex for Benign Brain Tumors (NausiCAA)
Acronym: NausiCAA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2024/14
Record Dates: First submitted 2024-06-19; First posted 2024-07-17 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Benign Brain Tumor
Keywords: Radiation induced nausea; Dorsal vagal complex; Brain tumors; Brainstem; Dosimetric constraint
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Irradiated patients: Patients irradiated for benign brain tumor, without chemotherapy
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — Radiation

SUMMARY:
Patients irradiated to the brain frequently experience nausea. The dorsal vagal complex (DVC) area is a specific brainstem zone and has been identified as likely responsible for nausea. Existing clinical studies show correlation between dose to the DVC and nausea, but they concern tumors of the airways and upper digestive tract, where there are many confounding factors.

The aim of this study is to establish a ling between radiation dose to the DVC and nausea. Defining a dose threshold to the DVC will allow radiation oncologists to optimize radiation dose distribution and reduce nausea in patients.

DETAILED DESCRIPTION:
Patients irradiated to the brain frequently experience nausea. The dorsal vagal complex (DVC) area is a specific brainstem zone and has been identified as likely responsible for nausea. Existing clinical studies show correlation between dose to the DVC and nausea, but they concern tumors of the airways and upper digestive tract, where there are many confounding factors.

A retrospective study was carried out a in the radiotherapy oncology department of Bordeaux University Hospital on 102 patients irradiated for a benign brain tumor. This study showed that DVC irradiation was significantly associated with the onset of nausea. However, this symptom alters the quality of life on a daily basis.

The objective of this prospective, multicenter, non-interventional study is to evaluate, using nausea validated questionnaires : Functional Living Index-Emesis (FLIE score), the correlation between DVC irradiation and nausea in benign brain tumors, at the end of radiotherapy, 1 month later and 3 months later. Fatigue associated with brain irradiation will also be studied with BFI (Brief Fatigue Inventory).

If there is an established link, a secondary dose constraint on this structure will be able to be proposed to reduce nausea in these radiotherapy indications.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* With benign brain tumor
* Irradiated with conventional fractionation (1,8-2Gy/fraction)

Exclusion Criteria:

* History of brain radiation
* History of head and neck radiation
* Demencia
* Concurrent chemotherapy
* Nausea at the time of inclusion
* Anti-nausea treatment : corticosteroids, metoclopramide, setrons, other

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients irradiated with conventional fractionation (1,8-2Gy/fraction) for benign brain tumor
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Functional Living Index-Emesis (FLIE score) | At inclusion, at day 35 of radiotherapy, at 1 and 3 months after completion of radiotherapy
  Validated score with 9 items of Likert scale concerning nausea

SECONDARY OUTCOMES:
Nausea grading | At inclusion, at day 35 of radiotherapy, at 1 and 3 months after completion of radiotherapy
  Common Terminology Criteria for Adverse Events (CTCAE) V5.0
Brief Fatigue Inventory (BFI) | At inclusion, at day 35 of radiotherapy, at 1 and 3 months after completion of radiotherapy
  Validated score with 9 items of Likert scale concerning fatigue
Dosimetric parameters of the Dorsal Vagal Complex | One day after completion of radiotherapy
  Mean Dose to the Dorsal Vagal Complex
Dosimetric parameters of the Braintem | One day after completion of radiotherapy
  Mean Dose to the Braintem

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU de Bordeaux, Service de Radiothérapie, Bordeaux
  - Hospices Civils de Lyon, Service d'Oncologie Radiothérapie - Hôpital Neurologique, Lyon
  - Institut de cancérologie Strasbourg Europe (ICANS), Service d'Oncologie Radiothérapie, Strasbourg

IPD SHARING:
Plan to Share IPD: No